CLINICAL TRIAL: NCT02536703
Title: LOTUS-CHINA: Safety and Efficacy of Lotus Valve For Transcatheter Aortic Valve Implantation In Patients With Severe Aortic Stenosis In Chinese Population
Brief Title: Safety and Efficacy of Lotus Valve For TAVI In Patients With Severe Aortic Stenosis In Chinese Population
Acronym: LOTUS-CHINA
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Principal Investigator, Jian'an Wang,MD,PhD, President of Second Affiliated Hospital, School of Medicine, Zhejiang University & Chief of Cardiology, Second Affiliated Hospital, School of Medicine, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAHZJU CT005
Record Dates: First submitted 2015-08-27; First posted 2015-09-01 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2015-08

CONDITIONS: Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lotus Valve System (Experimental): Transcatheter Aortic Valve Implantation (TAVI) with Lotus Valve System
  Interventions: Device: Lotus Valve System

INTERVENTIONS:
Device: Lotus Valve System — Lotus Valve System

SUMMARY:
To confirm the safety and efficacy of the Lotus™ Valve System in the Chinese population for Transcatheter Aortic Valve Implantation (TAVI) in symptomatic patients with severe aortic stenosis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with symptomatic severe aortic stenosis (echocardiographic criteria: AV effective orifice area (EOA) of < 1 cm2, mean AV gradient of > 40 mmHg, or AV peak systolic velocity of > 4.0 m/s; NYHA-class II or greater, angina pectoris, or syncope)
2. Subject has been informed of the nature of the study, agrees to its provisions and has provided written informed consent.
3. The subject agrees to comply with specified follow-up evaluations and to return to the investigational site where the procedure was performed.
4. Patients are technical and anatomical eligible for interventions

Exclusion Criteria:

1. A known hypersensitivity or contraindication to any of the following which cannot be adequately pre-medicated:

   Aspirin Heparin (HIT/HITTS) and bivalirudin Nitinol (titanium or nickel) Ticlopidine and clopidogrel Contrast media
2. Subject refuses a blood transfusion.
3. Other medical, social, or psychological conditions that in the opinion of an Investigator precludes the subject from appropriate consent.
4. Native aortic annulus size < 20 mm or > 29 mm per the baseline diagnostic imaging.
5. Life expectancy is less than one year

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-09; Primary Completion 2015-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Combined rate of death from any cause, myocardial infarction, and stroke | 30 days following procedure
  Outcome measures will be defined as suggested by the Valvular Academic Research Consortium (VARC)

SECONDARY OUTCOMES:
Number of participants with procedural complications | 30 days following procedure
Functional status (NYHA-classification) | 6 months following procedure
Echocardiographic prosthesis status | 6 months following procedure
Quality of Life (SF-12) | 6 months following procedure

CONTACTS AND LOCATIONS:
Overall Officials: Jian-an Wang, MD,PhD, Principal Investigator — Second Affiliated Hospital Zhejiang University School of Medicine
Locations (1):
- 2nd Affiliated Hospital, School of Medicine at Zhejiang University, Hangzhou, Zhejiang, China